CLINICAL TRIAL: NCT02349516
Title: A Randomized, Controlled Study of the Safety and Efficacy of Squalamine Lactate Eye Drops in Combination With Ranibizumab in Patients With Diabetic Macular Edema
Brief Title: Squalamine Lactate Eye Drops in Combination With Ranibizumab in Patients With Diabetic Macular Edema (DME)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled as of 9/12/15. 0 subjects enrolled.
Sponsor: Starr Muscle (Other)
Collaborators: Ohr Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor-Investigator, Starr Muscle, MD, primary investigator, Prism Vision Group
Organization: Prism Vision Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ohr-005
Record Dates: First submitted 2014-06-02; First posted 2015-01-29 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — squalamine lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Squalamine Solution BID 0.2% (Experimental): Squalamine Lactate Ophthalmic Solution 0.2% administered twice a day for 52 weeks in combination with monthly intravitreal injections of ranibizumab 0.3mg from baseline through week 20 and ranibizumab as needed from week 24 through week 52
  Interventions: Drug: Squalamine Lactate Ophthalmic Solution 0.2%
- Vehicle Solution 0.2% BID (Placebo Comparator): Vehicle Ophthalmic Solution 0.2% administered twice a day for 52 weeks in combination with monthly intravitreal injections of ranibizumab 0.3mg from baseline through week 20 and ranbizumab as needed from week 24 through week 52
  Interventions: Drug: Squalamine Lactate Ophthalmic Solution 0.2%
- Squalamine Solution 0.2% QID (Experimental): Squalamine Lactate Ophthalmic Solution 0.2% administered four times a day for 52 weeks in combination with monthly intravitreal injections of ranibizumab 0.3mg from baseline through week 20 and ranibizumab as needed from week 24 through week 52
  Interventions: Drug: Squalamine Lactate Ophthalmic Solution 0.2%
- Vehicle Solution 0.2% QID (Placebo Comparator): Vehicle Ophthalmic Solution 0.2% administered four times a day for 52 weeks in combination with monthly intravitreal injections of ranibizumab 0.3mg from baseline through week 20 and ranbizumab as needed from week 24 through week 52
  Interventions: Drug: Squalamine Lactate Ophthalmic Solution 0.2%

INTERVENTIONS:
Drug: Squalamine Lactate Ophthalmic Solution 0.2% — Squalamine Lactate Ophthalmic Solution 0.2% eye drop to be administered to study eye either BID or QID for 52 weeks
  Other Names: squalamine lactate

SUMMARY:
A randomized, controlled study of the safety and efficacy of Squalamine Lactate Eye Drops in combination with Ranibizumab intravitreal injections in patients with diabetic macular edema. The study duration is 52 weeks and patients will be randomized to one of four treatment arms.

DETAILED DESCRIPTION:
A randomized, controlled study of the safety and efficacy of Squalamine Lactate eye drops in combination with Ranibizumab intravitreal injections in patients with diabetic macular edema. Subjects will be randomized to one of the following treatment arms:

1. Squalamine Lactate Ophthalmic Solution administered twice a day for 52 weeks in combination with monthly injections of ranibizumab from baseline through week 20 and ranibizumab as needed from week 24 through week 52.
2. Vehicle Ophthalmic Solution administered twice a day for 52 weeks in combination with monthly injection of ranibizumab from baseline through week 20 and ranibizumab as needed from week 24 through week 52.
3. Squalamine Lactate Ophthalmic Solution administered four times a day for 52 weeks in combination with monthly injections of ranibizumab from baseline through week 20 and ranibizumab as needed from week 24 through week 52.
4. Vehicle Ophthalmic Solution administered four times a day for 52 weeks in combination with monthly injection of ranibizumab from baseline through week 20 and ranibizumab as needed from week 24 through week 52.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have clinically significant diabetic macular edema of ≥ 300 microns with central involvement using the Heidelberg or Cirrus machine
* Best corrected visual acuity of 20/32 to 20/320 inclusive in the study eye
* Adults ≥ 18 years of age with type 1 or 2 diabetes mellitus with diabetic macular edema

Exclusion Criteria:

* History of vitreoretinal surgery in the study eye
* Panretinal laser photocoagulation or macular laser photocoagulation in the study eye within 3 months of screening
* Any prior laser in study eye
* Previous use of intraocular or periocular corticosteroids in the study eye within 6 months of screening
* Previous treatment with anti-angiogenic drugs in either eye within 3 months of screening
* Uncontrolled diabetes mellitus with HbA1c levels greater than 12
* Ocular disorders in the study eye, other than diabetic macular edema, that my confound interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To explore the effect of Squalamine Lactate eye drops on Best Corrected Visual Acuity in subjects with diabetic macular edema | Mean change from baseline to Week 24
  Proportion of patients gaining at least 3,4 and 5 lines in best corrected visual acuity from baseline to week 24

SECONDARY OUTCOMES:
To assess the change in Central Retinal Thickness | Change at week 24 and at week 52
  Change in central retinal thickness at week 24 and at week 52
To assess need for rescue injections of Ranibizumab 0.3mg | Week 24 through week 52
  To assess the number of rescue (as needed) ranibizumab re-treatments from week 24 through week 52
To assess the safety and tolerability of Squalamine Eye Drops, measured by ophthalmic examination, the recording and evaluation of clinical AEs | At week 24 and at Week 52
  Ongoing safety assessments will include ophthalmic examination, the recording and evaluation of clinical AEs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — Prism Vision Group
Locations (1):
- NJ Retina, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Study cancelled, no data